CLINICAL TRIAL: NCT05768503
Title: Chidamide+Sintilimab+Bevacizumab Versus Standard Second-Line Therapy of FOLFIRI+Bevacizumab in Subjects With Advanced Microsatellite Stable (MSS/pMMR) Colorectal Cancer Who Have Failed Oxaliplatin-Containing First-Line Therapy
Brief Title: Comparing Chidamide+Sintilimab+Bev With Standard Second-line FOLFIRI+Bev in Advanced MSS/pMMR mCRC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, President, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPability-02
Record Dates: First submitted 2023-02-16; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Metastatic Microsatellite-stable Colorectal Cancer
Keywords: Colorectal Cancer; Microsatellite Stable; Chidamide; Sintilimab; PD-1; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drugs, Investigational; Tin Fluorides

STUDY DESIGN:
Intervention Model Description: 176 subjects will be randomized in a 1:1 ratio into either the chidamide + sintilimab + bevacizumab group or the standard second-line FOLFIRI + bevacizumab therapy group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chidamide + Sintilimab + Bevacizumab Group (Experimental): The treatment option for the chidamide + sintilimab + bevacizumab is 200 mg of sintilimab IV Drip Q3W, 30 mg of chidamide PO BIW, and bevacizumab 7.5 mg/kg IV Drip Q3W until loss of clinical benefit or development of intolerable toxicity (whichever occurs first), with a maximum treatment duration of 2 years.
  Interventions: Drug: Experimental drug
- FOLFIRI + Bevacizumab Group (Active Comparator): The treatment option for the standard second-line FOLFIRI + bevacizumab therapy group is bevacizumab 5 mg/kg IV Drip Q2W, irinotecan 180 mg/m2 IV Drip Q2W, calcium folinate 400 mg/m2 IV Q2W or calcium levofolinate 200 mg/m2 IV Drip Q2W, 5-fluorouracil 400 mg/m2 IV +2400 mg/m2 CIV (infusion 46-48 hr) Q2W until loss of clinical benefit or development of intolerable toxicity (whichever occurs first), with a maximum treatment duration of 2 years.
  Interventions: Drug: Control Rx

INTERVENTIONS:
Drug: Experimental drug — The treatment option for the chidamide + sintilimab + bevacizumab is 200 mg of sintilimab IV Drip Q3W, 30 mg of chidamide PO BIW, and bevacizumab 7.5 mg/kg IV Drip Q3W until loss of clinical benefit or development of intolerable toxicity (whichever occurs first), with a maximum treatment duration of 2 years.
  Other Names: CAP
  Arms: Chidamide + Sintilimab + Bevacizumab Group
Drug: Control Rx — The treatment option for the standard second-line FOLFIRI + bevacizumab therapy group is bevacizumab 5 mg/kg IV Drip Q2W, irinotecan 180 mg/m2 IV Drip Q2W, calcium folinate 400 mg/m2 IV Q2W or calcium levofolinate 200 mg/m2 IV Drip Q2W, 5-fluorouracil 400 mg/m2 IV +2400 mg/m2 CIV (infusion 46-48 hr) Q2W until loss of clinical benefit or development of intolerable toxicity (whichever occurs first), with a maximum treatment duration of 2 years.
  Other Names: FOLFIRI+BEV
  Arms: FOLFIRI + Bevacizumab Group

SUMMARY:
This is a randomized, controlled, multicenter phase Ⅲ study to evaluate the therapeutic efficacy and safety of chidamide + sintilimab + bevacizumab versus standard second-line FOLFIRI + bevacizumab therapy in subjects with advanced microsatellite stable colorectal cancer who have failed first-line oxaliplatin-containing standard therapy. The primary purpose is to compare the progression-free survival (PFS) of chidamide + sintilimab + bevacizumab versus standard second-line FOLFIRI + bevacizumab therapy for colorectal cancer, with a planned enrollment of 176 subjects with advanced microsatellite stable colorectal cancer who have failed first-line oxaliplatin-containing standard therapy.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio into either the chidamide + sintilimab + bevacizumab group or the standard second-line FOLFIRI + bevacizumab therapy group. The treatment option for the chidamide + sintilimab + bevacizumab (study group) is 200 mg of sintilimab IV Drip Q3W, 30 mg of chidamide PO BIW, and bevacizumab 7.5 mg/kg IV Drip Q3W, with a maximum treatment duration of 2 years. The treatment option for the standard second-line FOLFIRI + bevacizumab therapy group (control group) is bevacizumab 5 mg/kg IV Drip Q2W, irinotecan 180 mg/m2 IV Drip Q2W, calcium folinate 400 mg/m2 IV Q2W or calcium levofolinate 200 mg/m2 IV Drip Q2W, 5-fluorouracil 400 mg/m2 IV +2400 mg/m2 CIV Q2W, with a maximum treatment duration of 2 years.

The primary endpoint of this study is the progression-free survival (PFS), defined as the time from random assignment of the subject to disease progression or death from any cause.

All eligible patients will be randomly assigned to either the trial or control group in a 1:1 ratio based on the following stratification factors: Whether the primary focus is located in the right-sided colorectum; Whether bevacizumab has been administered in the first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced unresectable or metastatic colorectal adenocarcinoma (excluding mixed adenosquamous carcinoma and other pathological types) confirmed by pathological histology or cytology.
2. Diagnosis of pMMR confirmed by PCR for microsatellite stability (MSS) or low microsatellite instability (MSI-L), or by immunohistochemistry for DNA mismatch repair (MMR) proteins, including MLH1, MSH2, MSH6 and PMS2 protein expression, which result in no protein deletion.
3. Patients who have failed first-line oxaliplatin-containing standard therapy and have imaging evidence (e.g., CT scan) or clinical evidence (e.g., cytology report of new ascites or pleural effusion) of disease progression during or after treatment; patients whose intolerance of toxicity has led to discontinuation of first-line oxaliplatin-containing standard therapy may be enrolled; relapse within 180 days after the last dose of oxaliplatin-containing adjuvant therapy.
4. There is at least one measurable lesion according to RECIST v1.1.
5. ECOG PS score is in the range of 0~1.
6. Subjects who have signed a written informed consent form and who are able to comply with the visits and related procedures specified in the protocol.
7. Aged ≥ 18 years old and ≤ 75 years old.
8. Expected survival time ≥ 18 weeks.
9. Female subjects of childbearing age or male subjects whose sexual partners are at childbearing age are required to take effective contraception measures throughout the treatment period and for 6 months after the treatment (see section 4.3 of the protocol).
10. Subjects having adequate organ and bone marrow functions with laboratory test values within 7 days prior to enrollment meeting the following requirements (no blood components, cell growth factors, albumin, and other corrective therapy drugs are allowed to be given within the first 14 days of obtaining laboratory tests), as follows:

1) Blood routine: absolute neutrophil count (ANC) ≥ 1.5×109/L; platelet count (PLT) ≥ 100×109/L; hemoglobin level (HGB) ≥ 9.0 g/dL.

2) Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN in subjects without liver metastases, and ALT and AST ≤ 5.0 × ULN in subjects with liver metastases; serum albumin ≥ 25 g/L.

3) Renal function: serum creatinine (Cr) ≤ 1.5 x ULN. 4) Patients with routine urine results showing urine protein <2+ or routine urine testing showing urine protein ≥ 2+ at baseline should undergo 24-hour urine collection and 24-hour urine protein quantification < 1 g.

5) Coagulation function: international normalized ratio (INR) ≤ 1.5×ULN and activated partial thromboplastin time (APTT) ≤ 1.5×ULN.

Exclusion Criteria:

1. Prior exposure to any anti-PD-1 antibody, anti-PD-L1 antibody, HDAC inhibitor, or irinotecan.
2. Receiving any investigational drug within 4 weeks prior to the first dose of the study drug.
3. Concurrent participation in another interventional clinical study, except in an observational (non-interventional) clinical study or in the follow-up phase of an interventional study.
4. Receiving the last dose of antitumor therapy (chemotherapy, targeted therapy, tumor immunotherapy, or tumor embolization) within 3 weeks prior to the first dose.
5. Receiving radiotherapy within 4 weeks prior to the first dose.
6. Patients who have received radiotherapy more than 4 weeks prior to the first dose with any radiotherapy-related toxic reactions, such as radiation pneumonia, radiation hepatitis, radiation enteritis, including clinical symptoms only, or requiring glucocorticoid therapy.
7. Use of immunosuppressive drugs within 4 weeks prior to the first dose, excluding topical glucocorticoids by nasal spray, inhalation or other routes or physiological doses of systemic glucocorticoids (i.e., no more than 10 mg/day prednisone or equivalent doses of other glucocorticoids).
8. Receiving live attenuated vaccine within 4 weeks prior to the first dose or planning to receive during the study period.
9. Major surgical procedure (craniotomy, thoracotomy or open heart surgery) or unhealed wound, ulcer or fracture within 4 weeks prior to the first dose.
10. Presence of toxicity (excluding alopecia, non-clinically significant and asymptomatic laboratory abnormalities) from prior antineoplastic therapy not recovered to ≤ grade 1 by NCI common terminology criteriafor adverse events (CTCAE) Version 5.0 (NCI CTCAE Version 5.0) prior to the first dose.
11. Known presence of symptomatic CNS metastases and/or carcinomatous meningitis. Subjects with prior treatment for brain metastases may participate in the study provided that the brain metastases have remained stable for at least 4 weeks prior to the first dose of study treatment; and that neurological symptoms have recovered to ≤ grade 1 by NCI CTCAE version 5.0.
12. Active autoimmune disease requiring systemic therapy (e.g., use of disease-relieving drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are allowed. A known history of primary immunodeficiency. For patients with only positive autoimmune antibodies, the presence of autoimmune diseases should be confirmed at the discretion of the investigator.
13. Patients who are known to have active tuberculosis and are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year prior to the first dose.
14. Known to have interstitial lung disease requiring steroid hormone therapy.
15. Known to have acute or chronic active hepatitis B (HBsAg positive and HBV DNA ≥ 200 IU/mL or ≥ 103 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive).
16. Infected with human immunodeficiency virus (HIV) (HIV 1/2 antibody positive), known to be infected with syphilis.
17. Severe infections that are in the active phase or poorly controlled in clinical practice. Serious infection, including but not limited to hospitalization for complications of infection, bacteremia or severe pneumonia, within 4 weeks prior to the first dose.
18. Significant malnutrition, such as the need for intravenous supplemental nutrient solutions; except for malnutrition corrected more than 4 weeks prior to the first dose.
19. Symptomatic congestive heart failure (New York Heart Association class II-IV); symptomatic or poorly controlled arrhythmias.
20. Uncontrolled arterial hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) even with standard treatment.
21. Any arterial thromboembolic event including myocardial infarction, pulmonary embolism, and unstable angina within 6 months prior to enrollment.
22. A history of deep vein thrombosis or any other serious thromboembolism (implantable IV port or catheter-derived thrombosis, or superficial vein thrombosis is not considered "serious" thromboembolism) within 3 months prior to enrollment.
23. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B or more severe cirrhosis.
24. A history of gastrointestinal perforation and/or fistula in the previous 6 months; a history of peptic ulcer, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection complicated by chronic diarrhea), Crohn's disease, ulcerative colitis, abdominal abscess, or long-term chronic diarrhea. Post-intestinal stent implantation.
25. > 3 loose stools per day at baseline, suggesting a predisposition to colon or small bowel disease with uncontrollable symptoms.
26. A history of allergy or known intolerance to atropine sulfate or loperamide or the appropriate antiemetic in combination with FOLFIRI.
27. Uncontrolled metabolic disorders or other non-malignant organ or systemic diseases or secondary reactions to cancer and can lead to higher medical risk and/or uncertainty in survival evaluation.
28. A known history of inherited bleeding tendency disorders or coagulation disorders
29. Any life-threatening bleeding event within the previous 3 months, including the need for blood transfusion therapy, surgical or local treatment, or ongoing drug therapy.
30. A high risk of bleeding as determined by the investigators: cirrhosis with severe esophagogastric fundic varices, intermittent or persistent non-fatal bleeding events (including but not limited to intermittent bloody stools or positive occult blood due to primary intestinal lesions, intermittent hemoptysis due to pulmonary metastases).
31. Cerebrovascular accident (including transient ischemic attack) in the previous 6 months.
32. Use of aspirin (>325 mg/day) or other NSAIDs known to inhibit platelet function for 10 consecutive days within 10 days prior to the first dose.
33. Treatment with oral or parenteral anticoagulants or thrombolytics for 10 consecutive days within 10 days prior to the first dose. However, prophylactic use of anticoagulants is allowed.
34. Pleural fluid, ascites, and pericardial effusion with clinical symptoms or requiring drainage, except for small amounts of pleural fluid, small amounts of ascites, and small amounts of pericardial effusion without clinical symptoms on imaging only.
35. A history of other primary malignancies, except: malignancies in complete response for at least 2 years prior to enrollment and requiring no other treatment during the study period; adequately treated non-melanoma skin cancer or malignant freckled nevus with no evidence of disease recurrence; adequately treated carcinoma in situ with no evidence of disease recurrence.
36. A known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
37. Known to be allergic to any monoclonal antibody component.
38. Female subjects in the pregnancy or lactating period.
39. A history of alcohol or drug abuse.
40. Other acute or chronic illnesses, psychiatric disorders, or abnormal laboratory test values that may result in the following outcomes: increasing the risk associated with study participation or study drug administration, or interfering with the interpretation of study results and, at the investigator's discretion, classifying the patient as ineligible for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Around 4 years
  Time from randomization to disease progression or death from any cause

SECONDARY OUTCOMES:
Objective Response Rates (ORR) | Around 4 years
  The percentage of subjects whose therapeutic effect evaluation is complete response (CR) or partial response (PR) according to RECIST 1.1.
Overall Survival (OS) | Around 4 years
  Time from randomization to death from any cause
Disease Control Rate (DCR) | Around 4 years
  The percentage of subjects whose therapeutic effect evaluation is complete response (CR), partial response (PR) or stable disease (SD) according to RECIST 1.1.
Duration of Response (DOR) | Around 4 years
  Time from achievement of a response to disease progression.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) | Around 4 years
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, Tumor Assessment Visit (Week 8 and 12) and End of Treatment visit. The higher score means the worse quality of life.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CR29 (EORTC QLQ-CR29) | Around 4 years
  Quality of life in patients with colorectal cancer is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) CR29. It will be evaluated at Screening, Tumor Assessment Visit (Week 8 and 12) and End of Treatment visit. The higher score means the worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (12):
- China (12):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No